CLINICAL TRIAL: NCT01904513
Title: Investigating the Effects of Probiotic Yogurt on Reducing the Levels of Environmental Toxins Among School Children in Mwanza, Tanzania
Acronym: PDTX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Principal Investigator, Dr. Gregor Reid, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 102881
Record Dates: First submitted 2013-07-04; First posted 2013-07-22 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: C535854; D004786
Keywords: Metals; Pesticides; Toxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Daily consumption of yogurt supplemented with L. rhamnosus GR-1 at ~10^10 CFU/day
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GR-1
- Milk (Other): Daily consumption of pasteurized whole milk
  Interventions: Dietary Supplement: Pasteurized Whole Milk

INTERVENTIONS:
Dietary Supplement: Pasteurized Whole Milk
  Arms: Milk
Dietary Supplement: Lactobacillus rhamnosus GR-1
  Other Names: L. rhamnosus ATCC 55826
  Arms: Probiotic

SUMMARY:
The primary objective of this pilot study is to determine if consumption of a probiotic yogurt causes reduced levels of environmental toxins in a group of school-aged Tanzanian children. The secondary objective is to determine the levels of environmental toxins in Tanzanian children and compare these to literature values of levels believed to negatively affect health and development. The third objective is to analyze the intestinal microbiota of the children and to determine if consumption of a probiotic yogurt has a significant affect on the microbiota composition.

DETAILED DESCRIPTION:
A group of 60 first year students from the Lake Primary School will be recruited for inclusion into the study. After gaining consent from the child's caregiver, each child will be given a participant number and blood, urine and fecal samples will be collected from each child by qualified personnel from NIMR. Children will be randomized into two groups (n=30) to match age, sex and weight, one of which will receive a 100 g probiotic yogurt containing Lactobacillus rhamnosus GR-1 while the other group will receive an equivalent portion of milk. After 30 days of consuming the yogurt or milk, samples will again be collected.

Samples will be shipped back to London, Ontario Canada on dry ice for analysis. Blood and urine will be analyzed via high-resolution sector field inductively coupled plasma mass spectrometry (HR-SF-ICP-MS) to determine levels of toxic heavy metals (Mercury, Lead, Cadmium, Arsenic). This will be carried out by the London Health Sciences Trace Elements laboratory in Canada. Urine will also be analyzed via gas chromatography/ mass spectrometry (GC-MS) to determine levels of pesticides at the Biotron Facility (University of Western Ontario). We will also examine urine via NMR for potential host metabolic changes in response to probiotic instillation.

Bacterial community DNA samples will be extracted and analyzed to determine the gastrointestinal microbiota of the children both before and after administration of the probiotic yogurt to determine the effect of the yogurt on the gut microbiome. Briefly, DNA will be extracted with the Qiagen Stool DNA extraction kit and bacterial community 16S rRNA genes will amplified using barcoded primers specific for a variable region within the gene. The samples will be pooled and sequenced on the Ion Torrent platform (London Regional Genomics Center, Canada). Reads are then processed and analyzed using custom scripts as well as the Quantitative Insights Into Microbial Ecology (QIIME) tool, which is the leading package for microbiota analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-10
* Attends Lake Primary School (Mwanza, Tanzania)

Exclusion Criteria:

* Allergic to milk/ milk products
* Lactose intolerant

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes in Body Toxin Levels | Before and after the 25 day intervention period.
  Body toxin levels (metals, pesticides) by HR-SF-ICP-MS and GC/MS.

SECONDARY OUTCOMES:
Changes in Microbiota Composition | Before and after the 25 day intervention period.
  Stool microbiota composition shifts as determined by 16S rRNA profiling.
Microbes linked to host toxin levels | Initial sample collection visit
  Microbes, as determined via 16S rRNA sequencing, associated with high toxin levels.
Changes in host metabolism due to probiotic instillation | Before and after the 25 day intervention period.
  Host metabolic shifts as measured by NMR from urine

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute for Medical Research, Mwanza, Tanzania

REFERENCES:
- [Derived] Bisanz JE, Enos MK, Mwanga JR, Changalucha J, Burton JP, Gloor GB, Reid G. Randomized open-label pilot study of the influence of probiotics and the gut microbiome on toxic metal levels in Tanzanian pregnant women and school children. mBio. 2014 Oct 7;5(5):e01580-14. doi: 10.1128/mBio.01580-14. PMID 25293764